CLINICAL TRIAL: NCT04193644
Title: Effects of Various Types of Physical Activity on Tumor-specific Symptoms of Fatigue in Breast Cancer Patients Undergoing Chemotherapy and / or Radiotherapy
Brief Title: Mindfulness and Self-compassion Focussed Walking
Acronym: MSCW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sana-Klinikum Lichtenberg (Other); Park-Klinik Berlin Weißensee (Unknown); Vivantes Klinikum am Urban (Unknown); Steffen Lohrer Stiftung (Unknown)
Responsible Party: Principal Investigator, Yves Steininger, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSCW2019
Record Dates: First submitted 2019-11-30; First posted 2019-12-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Fatigue
Keywords: tumor-specific fatigue syndrome; mindfulness; self-compassion
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking-Group (Active Comparator): Participants in this group walk 45 minutes 3 times a week (plus 15 minutes of warm up and cool-down) in a moderate intensity range (64-76% HRmax).
  Interventions: Behavioral: Walking training
- Mindfulness and Self-Compassion focussed Walking-Group (Experimental): Participants in this group walk 45 minutes 3 times a week (plus 15 minutes of warm up and cool-down) in a moderate intensity range (64-76% HRmax) and additionally practice mindfulness exercises and self-compassion exercises during the 60 minutes.
  Interventions: Behavioral: Mindfulness and Self-Compassion focussed exercises during walking training
- TAU-Group (No Intervention): Participants in this group receive no intervention.

INTERVENTIONS:
Behavioral: Mindfulness and Self-Compassion focussed exercises during walking training — Mindfulness and Self-Compassion focussed exercises during walking training with moderate intensity
  Arms: Mindfulness and Self-Compassion focussed Walking-Group
Behavioral: Walking training — Walking training with moderate intensity
  Arms: Walking-Group

SUMMARY:
This research study is evaluating the effects of two training programs (1. Walking, 2. Mindfulness and Self-compassion focussed Walking) on tumor-specific symptoms of fatigue in women with breast cancer undergoing chemo- and/or radiotherapy.

DETAILED DESCRIPTION:
This randomized research study is evaluating the effects of two training programs (1. Walking, 2. Mindfulness and Self-compassion focussed Walking (MSCW)) on tumor-specific symptoms of fatigue in women with breast cancer undergoing chemo- and/or radiotherapy. The results of both groups are compared with each other and with those of a control group.

The MSCW program combines endurance based physical activity in the form of medically controlled walking, as well as standardized, evidence-based mindfulness exercise elements in a training program.

The participants of both active groups (Walking and MSCW) practice for 12 weeks, once a week for 60 minutes under the guidance of a trainer in a group and 2 additional times (60 minutes each) independently at home.

The purpose of this study is to prevent a sharp decline in quality of life due to fatigue symptoms by participating in the MSCW training program.

A total of 135 participants will be included in the study. All participants are followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer who have started antineoplastic therapy (chemotherapy / radiotherapy).
* Age ≥18 years
* The patient must be able to perform the study intervention (physically and psychologically).
* oral and written consent to participate in the study.

Exclusion Criteria:

* distant metastases
* Severe mental and / or additional organic illnesses
* Clinically relevant cardiac arrhythmias or angina pectoris
* Severe pulmonary disease
* inadequate walking ability or gait disturbance (including neurological deficits, endoprosthesis supply that lead to gait insecurity)
* regular meditation practice (several times a week)
* Planned start of meditation, relaxation, MBSR, yoga, Qi Gong courses over the next 24 weeks.
* Participation in other intervention studies on walking or meditation
* Insufficient knowledge of the German language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor specific fatigue symptomatology | Change from baseline to 12, 24 and 52 weeks
  Fatigue Assessment Questionnaire (FAQ), minimum value 0, maximum value 60, higher values mean a worse outcome

SECONDARY OUTCOMES:
Disease-specific quality of life | Change from baseline to 12, 24 and 52 weeks
  Functional Assessment of Cancer Therapy - Breastcancer (FACT-B), minimum value 0, maximum value 148 for FACT-B total score, minimum value 0, maximum value 28 for subscores, higher values mean a better outcome
Self-Compassion | Change from baseline to 6, 12, 24 and 52 weeks
  Self-Compassion Scale German (SCS-D), minimum value 1, maximum value 5 for SCS-D total score, minimum value 1, maximum value 5 for subscores, higher values mean a better outcome
Mindfulness | Change from baseline to 6, 12, 24 and 52 weeks
  Southampton Mindfulness Questionnaire (SMQ), minimum value 0, maximum value 96 for SMQ total score, minimum value 0, maximum value 24 for subscores, higher values mean a better outcome
Anxiety and depression | Change from baseline to 12, 24 and 52 weeks
  Hospital Anxiety and Depression Scale (HADS), minimum value 0, maximum value 42 for HADS total score, minimum value 0, maximum value 21 for subscores, higher values mean a worse outcome
Stress | Change from baseline to 12, 24 and 52 weeks
  Perceived Stress Scale (PSS), minimum value 0, maximum value 40 for PSS total score, higher values mean a worse outcome
Anxiety | Change from baseline to 12, 24 and 52 weeks
  State-Trait Anxiety Inventory (STAI) - Trait Dimension, minimum value 10, maximum value 80 for STAI total score, higher values mean a better outcome
Heart rate variability | Change from baseline to 12, 24 and 52 weeks
  Polar watch V800
Alpha-Amylase | Change from baseline to 12, 24 and 52 weeks
  extraction from saliva measurements
cardiac function parameters | Change from baseline to 12, 24 and 52 weeks
  Examination by sonography
Immune defence | Change from baseline to 12, 24 and 52 weeks
  Measurement of leukocytes by blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof., Study Director — Charite Universitätsmedizin Berlin
Locations (2):
- Germany (2):
  - Charite Universitätsmedizin Berlin, Berlin
  - Sana-Klinikum Lichtenberg, Berlin, Berlin